CLINICAL TRIAL: NCT03033407
Title: A Randomized, Controlled, Open-label Study to Evaluate the Efficacy of the S-Diabetes Care Program Based on Ubiquitous Healthcare System in Patients With Type 2 Diabetes
Brief Title: A Study to Evaluate the Efficacy of Diabetes Management Based on Ubiquitous Healthcare System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kangbuk Samsung Hospital (Other)
Responsible Party: Principal Investigator, Cheol-Young Park, Prof., Kangbuk Samsung Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: KBSMC 2014-09-021
Record Dates: First submitted 2017-01-18; First posted 2017-01-26 (Estimated); Last update posted 2017-01-26 (Estimated); Status verified 2017-01

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Masking Description: It was open label study.

ARMS (2):
- Intervention-Maintenance group (Experimental): Intervention was adding 'Tailored mobile coaching messages' onto conventional diabetes management. This study was divided into two phases. In six-month phase 1 study, the participants in I-M group received tailored mobile coaching. And during the second half six-month phase 2 study, they could receive only regular information messages without individualized coaching.
  Interventions: Other: Tailored mobile coaching messages
- Control-Intervention group (Active Comparator): Intervention was adding 'Tailored mobile coaching messages' onto conventional diabetes management. In six-month phase 1 study, the participants in Control-Intervention group maintained usual care for diabetes. During the second half six-month phase 2 study, they received tailored mobile coaching.
  Interventions: Other: Tailored mobile coaching messages

INTERVENTIONS:
Other: Tailored mobile coaching messages — Intervention was adding tailored mobile coaching to current usual diabetes care. The participants received regular mobile messages via Switch app according to entered data, such as self-monitoring of blood glucose, blood pressure, exercise, dietary record, medication record, and body weight. Contents of messages were alert for the unused, weather, behavioral recommendation, education about diabetes, and individualized advices.

SUMMARY:
The aim of this study is to investigate whether adding tailored mobile coaching system to present community primary care for diabetes management would result in better glycemic control and other diabetes-related outcomes in adult patients with type 2 diabetes, compared with maintaining usual diabetes management only.

DETAILED DESCRIPTION:
The incidence and prevalence of type 2 diabetes is increasing rapidly worldwide. Considering the fact that complications of diabetes result in greater expenditure and reduced productivity is a socioeconomic concern, adequate glycemic control is important not only as individual health problem but also as challenge to healthcare systems worldwide. To support patients' behavior change efforts, including healthy lifestyle choices, disease self-management, and prevention of diabetes complication, multifaceted professional interventions are needed. Ubiquitous healthcare based on information and communication technology is one of these approaches.

The aim of this study is to investigate whether adding tailored mobile coaching system to present community primary care for diabetes management would result in better glycemic control and other diabetes-related outcomes in adult patients with type 2 diabetes, compared with maintaining usual diabetes management only.

ELIGIBILITY:
Inclusion Criteria:

* Korean policyholders with type 2 diabetes;
* Aged ≥ 19 years;
* Smartphone users;
* Glycated hemoglobin (HbA1c) ≥ 6.5% within 3 months.

Exclusion Criteria:

* Currently had serious concomitant disease other than diabetes;
* Had admission histories due to malignancy, myocardial infarction, cerebral infarction, or organ transplantation;
* Pregnant or had plan for pregnancy within 6 months;
* Planned for attending other clinical;
* Illiteracy.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2014-10; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
glycated hemoglobin levels | at 6 months

SECONDARY OUTCOMES:
change in glycated hemoglobin levels within each group | between baseline and 6 months
change in body mass index within each group | between baseline and 6 months
change in low-density lipoprotein cholesterol within each group | between baseline and 6 months
change in high-density lipoprotein cholesterol within each group | between baseline and 6 months
change in triglyceride within each group | between baseline and 6 months
change in blood pressure within each group | between baseline and 6 months

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lee MK, Lee DY, Ahn HY, Park CY. A Novel User Utility Score for Diabetes Management Using Tailored Mobile Coaching: Secondary Analysis of a Randomized Controlled Trial. JMIR Mhealth Uhealth. 2021 Feb 24;9(2):e17573. doi: 10.2196/17573. PMID 33625363